CLINICAL TRIAL: NCT03615690
Title: The Influence of a Fasting Mimicking Diet on Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sidhartha Ranjit Sinha, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 47075
Record Dates: First submitted 2018-07-03; First posted 2018-08-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Disease; Diet Modification; Ulcerative Colitis
Keywords: ulcerative colitis; IBD; diet; fasting; fasting mimicking diet; UC; intermittent fasting
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Fasting; Intermittent Fasting | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting Mimicking Diet (Experimental): Three cycles of a 5-day reduced calorie diet
  Interventions: Other: Fasting Mimicking Diet
- Regular Diet Control Arm (Placebo Comparator)
  Interventions: Other: Regular Diet

INTERVENTIONS:
Other: Fasting Mimicking Diet — 5 day reduced calorie diet
  Arms: Fasting Mimicking Diet
Other: Regular Diet — Regular Diet
  Arms: Regular Diet Control Arm

SUMMARY:
The purpose of this study is to see how a diet that mimics fasting effects inflammation in patients with mild to moderate Ulcerative Colitis (UC). The diet may allow users to receive the benefits of fasting while also being able to enjoy food (the ingredients of which are GRAS (generally recognized as safe) by the Food and Drug Administration (FDA). Research on dietary interventions and UC are very limited. Fasting mimicking diets (FMD) have been studied with support of the National Institute of Health and published in leading journals. This research investigates whether markers of inflammation decrease and/or quality of life increases after three cycles of a five-day period of the fasting mimicking diet, and may provide rationale for its use to treat UC.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Ulcerative Colitis on the partial Mayo Score out of 9 (score between 2 to 7)
* Age of 18-70 at start of study (inclusive)

Exclusion Criteria:

* Women who are pregnant or nursing or expect to be pregnant
* Individuals allergic to nuts
* Individuals with a body mass index (BMI) lower than 18
* Individuals diagnosed with a serious medical condition as defined by the patient's physician, unless approved in writing by a physician
* Individuals who have been severely weakened by a disease or medical procedure,
* Individuals who are taking medication which may not be safely consumed with a calorie restricted diet
* Individuals with diabetes who are taking anti-diabetic drugs associated with risk of hypoglycemia
* Individuals with more than mild-moderate cardiovascular disease or life-threatening cancer (as determined by patient's physician) unless approved by a physician
* Individuals with history of severe cardiac disease (particularly uncompensated congestive heart failure NYHA grade 2 or more or LVEF < 40%)
* Individuals with a history of syncope
* Individuals with dietary needs incompatible with the FMD meal plan
* Individuals with liver or kidney disorders that may be affected by very low glucose and protein content of the diet.
* Patients on a caloric restricted diet will also be excluded.
* Patients with relevant prior gastrointestinal surgery and consequences such as short bowel syndrome, ostomy of small or large intestine, hemi- or total colectomy, proctocolectomy, ileoanal pouch will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical response as per partial Mayo score | Comparison of disease score up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as a decrease from baseline in the partial Mayo score of >= 2 points and either a rectal bleeding subscore of <=1 or a decrease in the rectal bleeding subscore of >=1 point, or achieving a partial Mayo score <2. The partial Mayo score consists of the subscores for stool frequency, rectal bleeding, and PGA, omitting endoscopy.

SECONDARY OUTCOMES:
Clinical remission as per partial Mayo score | Comparison of disease score up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as a partial Mayo score < 2 points. The partial Mayo score consists of the subscores for stool frequency, rectal bleeding, and PGA, omitting endoscopy.
Clinical remission as per modified Mayo (mMayo) score | Comparison of disease score up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as mMayo score <= 1 point, with rectal bleeding and stool frequency subscore of 0, and endoscopy subscore of 0 or 1. The mMayo score consists of the subscores for stool frequency, rectal bleeding, and endoscopy, omitting PGA.
Clinical response as per mMayo score | Comparison of disease score up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as a decrease of the mMayo score of >=2 points and either a rectal bleeding subscore of <=1 or a decrease in the rectal bleeding subscore of >=1 point.
Patient global assessment | Assessed within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  "Do you believe you are in remission from your UC symptoms?" (Yes/No). No scale.
Change in C-Reactive Protein (CRP). | Comparison of CRP levels up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Change in the inflammatory marker CRP (if elevated at baseline).
Change in Erythrocyte Sedimentation Rate (ESR). | Comparison of ESR levels up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Change of the inflammatory marker ESR (if elevated at baseline).
Change in Fecal Calprotectin. | Comparison of calprotectin levels up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Change of the inflammatory marker fecal calprotectin (if elevated at baseline).
Effect of FMD on endoscopic outcomes | Comparison of disease score up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Changes in modified Mayo (mMayo) endoscopic subscore. The subscore ranges from 0 to 3 points with higher scores reflecting more severe disease.
Symptomatic remission as per Patient Reported Outcome (PRO2) score | Comparison of disease score up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as a Mayo stool frequency subscore of 0 or 1 and a Mayo rectal bleeding subscore of 0.
Change in Short Inflammatory Bowel Disease questionnaire (SIBDQ) score | Comparison of SIBDQ score up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Quality of life score in UC patients. Response to each of the questions is graded from 1 to 7 (1 being the worst situation and 7 the best).

OTHER OUTCOMES:
Assessment of primary and key secondary endpoints at baseline versus 3 months after the start of Cycle 3. | Comparison of endpoints up to 14 days before starting Cycle 1, and 3 months after the start of Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Outcomes 1 to 11 at additional time points.
Changes in cytokines/chemokines and immune cell profiles using flow cytometry and mass cytometry (CyTOF). | Comparison of cytokines/chemokines/immune cell profiles up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Cytokines/chemokines (e.g. TNF-alpha, IL-6, IL-10, IFN-gamma, α4β7, CCR1, and CCR9) and immune cell profiles.
Differences in clinical markers of disease activity at baseline versus within 6 days after completing Cycle 1. | Comparison of clinical markers up to 14 days before starting Cycle 1, and within 6 days after completing Cycle 1. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Clinical markers of disease activity are CRP, ESR and fecal Calprotectin (if elevated at baseline).
Changes in gut metabolites (including short-chain fatty acid and bile acid profiles) and microbiome profiles (using 16S rRNA/shotgun metagenomics). | Comparison of characteristics up to 14 days before Cycle 1, within 6 days after completing Cycle 3, and 3 months after start of Cycle 3. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Gut metabolites include short-chain fatty acid and bile acid profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Sidhartha R Sinha, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States